CLINICAL TRIAL: NCT04962230
Title: A PHASE 1, OPEN-LABEL, FIXED SEQUENCE, 2-PERIOD CROSSOVER STUDY TO ESTIMATE THE EFFECT OF CARBAMAZEPINE ON THE PHARMACOKINETICS OF PF-07321332 BOOSTED WITH RITONAVIR IN HEALTHY PARTICIPANTS
Brief Title: Drug-Drug Interaction Study Assessing Effect of Carbamazepine on PF-07321332 Boosted With Ritonavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: C4671014
Record Dates: First submitted 2021-07-10; First posted 2021-07-14 (Actual); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Healthy Participant
Keywords: Drug-drug interaction; Carbamazepine; CYP3A4 inducer
MeSH Terms: interventions — nirmatrelvir and ritonavir drug combination; Carbamazepine; Ritonavir

STUDY DESIGN:
Intervention Model Description: This is a Phase 1, fixed sequence, 2-period study to estimate the effect of a strong CYP3A4 inducer, carbamazepine, on the PK of PF-07321332 and ritonavir in healthy participants. A total of approximately 12 healthy male and/or female participants will be enrolled into the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Period 1 (Experimental): PF-07321332/ritonavir orally as a single dose
  Interventions: Drug: PF-07321332/ritonavir
- Period 2 (Experimental): Carbamazepine + PF-07321332/ritonavir orally.
  Interventions: Drug: Carbamazepine; Drug: PF 07321332/ritonavir

INTERVENTIONS:
Drug: PF-07321332/ritonavir — PF-07321332/ritonavir administered orally as a single dose on Day 1, Period 1
  Arms: Period 1
Drug: Carbamazepine — In Period 2, Days 1-3, participants will receive low-dose of carbamazepine twice daily (BID), then a titrated mid-dose of carbamazepine BID on Days 4-7, and finally maintaining carbamazepine at the high-dose on Days 8-15.
  Arms: Period 2
Drug: PF 07321332/ritonavir — In Period 2, Day 14, participants will receive a single dose of PF-07321332/ritonavir orally.
  Arms: Period 2

SUMMARY:
This is a drug-drug interaction study to assess the effects of a single dose of PF-07321332/ritonavir after multiple dose administrations of carbamazepine. Pharmacokinetic (PK) will be evaluated for PF-07321332 and ritonavir. Carbamazepine is being utilized as a cytochrome P450 3A4 (CYP3A4) inducer.

ELIGIBILITY:
Inclusion Criteria:

1. Female participants of childbearing potential must have a negative (urine or serum) pregnancy test.
2. Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

1. Positive test reverse-transcriptase polymerase chain reaction (RT-PCR) result for SARS-CoV-2 infection at the time of Screening or Day -1.
2. Subjects shown to carry or be positive for human leukocyte antigen (HLA)-B*1502 and HLA-A*3101
3. Participants taking monoamine oxidase inhibitors (MAOIs) should discontinue MAOI for a minimum of 14 days prior to dosing in the current study.
4. Hormonal methods of contraception (including oral and transdermal contraceptives, injectable progesterone, vaginal ring, and postcoital contraceptive methods) and hormone replacement therapy must have been discontinued at least 28 days prior to the first dose of investigational product. Depo Provera must be discontinued at least 6 months prior to the first dose of study treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-10-09 (Actual); Study Completion 2021-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Background] Andreasen AH, Brosen K, Damkier P. A comparative pharmacokinetic study in healthy volunteers of the effect of carbamazepine and oxcarbazepine on cyp3a4. Epilepsia. 2007 Mar;48(3):490-6. doi: 10.1111/j.1528-1167.2007.00924.x. PMID 17346248
- [Result] Hsu A, Granneman GR, Bertz RJ. Ritonavir. Clinical pharmacokinetics and interactions with other anti-HIV agents. Clin Pharmacokinet. 1998 Oct;35(4):275-91. doi: 10.2165/00003088-199835040-00002. PMID 9812178
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4671014

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consisted of 2 periods. Twelve participants were enrolled into the study. All 12 participants were treated and 10 completed the study. Two participants discontinued from the study in Period 2.
Groups:
- All Participants: All participants were enrolled and received study drug. In Period 1, participants received PF-07321332 300 mg with ritonavir 100 mg administered orally as a single dose starting at approximately 0800 hours (±2 hours) on Day 1 following an overnight fast of at least 10 hours. PF-07321332 and ritonavir were dosed simultaneously (within no more than 5 minutes of each other). In Period 2, participants received carbamazepine 100 mg twice daily (BID) administered orally on Days 1, 2, and 3, and titrated up to 200 mg BID on Days 4, 5, 6, and 7, and eventually titrated up to and maintained at 300 mg BID stably in the rest of Period 2 from Days 8 to 15. Carbamazepine was administered with or without food on all study days except on Study Day 14 when dosing was under fasting conditions. There were no water restrictions for carbamazepine dosing. On Period 2 Day 14, participants received PF-07321332 300 mg administered orally with ritonavir 100 mg starting at approximately 0815 to 0830 hours (±10 minutes), approximately 15 to 30 min after the carbamazepine dose. PF-07321332 and ritonavir were dosed simultaneously (within no more than 5 minutes of each other).
Period: PF-07321332 300 mg/Ritonavir 100 mg
Arm/Group | All Participants
Started | 12
Completed | 12
Not Completed | 0
Period: Carbamazepine+PF-07321332/Ritonavir
Arm/Group | All Participants
Started | 12
Completed | 10
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: All participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Customized [Count of Participants; unit: Participants]
  Less than 18 years old （<18) | 0
  18 to 25 years old (18-25) | 1
  26 to 35 years old (26-35) | 4
  36 to 45 years old (36-45) | 2
  more than 45 years old （>45） | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 7
  More than one race | 1
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 9

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of PF-07321332
Description: Cmax was defined as maximum observed plasma concentration and can be observed directly from data.
Time Frame: Day 1 pre-dose, and at 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, and 48 hours post dose in Period 1; Day 14 pre-dose, and at 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, and 48 hours post-dose or early termination/discontinuation in Period 2
Population: The analysis population was defined as all participants assigned to investigational product and treated who had at least 1 of the PK parameters of primary interest measured. Number of participants analyzed represents the number of participants contributing to the summary statistics for Cmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Period1: PF-07321332 300 mg/Ritonavir 100 mg: In Period 1, participants received PF-07321332 300 mg with ritonavir 100 mg administered orally as a single dose starting at approximately 0800 hours (±2 hours) on Day 1 following an overnight fast of at least 10 hours. PF-07321332 and ritonavir were dosed simultaneously (within no more than 5 minutes of each other).
- Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg: In Period 2, participants received carbamazepine 100 mg BID administered orally on Days 1, 2, and 3, and titrated up to 200 mg BID on Days 4, 5, 6, and 7, and eventually titrated up to and maintained at 300 mg BID stably in the rest of Period 2 from Days 8 to 15. Carbamazepine was administered with or without food on all study days except on Study Day 14 when dosing was under fasting conditions. There were no water restrictions for carbamazepine dosing. On Period 2 Day 14, participants received PF-07321332 300 mg administered orally with ritonavir 100 mg starting at approximately 0815 to 0830 hours (±10 minutes) approximately 15 to 30 min after the carbamazepine dose. PF-07321332 and ritonavir were dosed simultaneously (within no more than 5 minutes of each other).
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
Number analyzed (Participants) | 12 | 10
nanogram per milliliter (ng/mL) | 2210 (33) | 1300 (43)
Statistical Analysis 1: Comparison: Period1: PF-07321332 300 mg/Ritonavir 100 mg vs Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg; Test type: Other — PF-07321332/ritonavir administered alone was the Reference treatment and PF-07321332/ritonavir coadministered with carbamazepine was the Test treatment; p = 0.05, Mixed Models Analysis; specify in comments = 56.82, 90% CI 2-sided [47.04 to 68.62] — Mixed Model was fitted to obtain: 1.Ratio of adjusted geometric means 2.90% CI for the ratios

2. Primary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of PF-07321332
Description: AUCinf was defined as area under the concentration-time curve from time 0 to infinity and was calculated as AUClast + (Clast*/kel), where Clast* is the predicted plasma concentration at the last quantifiable time point estimated from the log-linear regression analysis.
Time Frame: as for outcome 1
Population: The analysis population was defined as all participants assigned to investigational product and treated who had at least 1 of the PK parameters of primary interest measured. Number of participants analyzed represents the number of participants contributing to the summary statistics for AUCinf.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Period1: PF-07321332 300 mg/Ritonavir 100 mg: In Period 1, participants received PF-07321332 300 mg with ritonavir 100 mg administered orally as a single dose starting at approximately 0800 hours (±2 hours) on Day 1 following an overnight fast of at least 10 hours. PF 07321332 and ritonavir were dosed simultaneously (within no more than 5 minutes of each other).
- Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg: In Period 2, participants received carbamazepine 100 mg BID administered orally on Days 1, 2, and 3, and titrated up to 200 mg BID on Days 4, 5, 6, and 7, and eventually titrated up to and maintained at 300 mg BID stably in the rest of Period 2 from Days 8 to 15. Carbamazepine was administered with or without food on all study days except on Study Day 14 when dosing was under fasting conditions. There were no water restrictions for carbamazepine dosing. On Period 2 Day 14, participants received PF-07321332 300 mg administered orally with ritonavir 100 mg starting at approximately 0815 to 0830 hours (±10 minutes) approximately 15 to 30 min after the carbamazepine dose. PF 07321332 and ritonavir were dosed simultaneously (within no more than 5 minutes of each other).
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
Number analyzed (Participants) | 12 | 10
nanogram*hour per milliliter (ng*hr/mL) | 23010 (23) | 10280 (58)
Statistical Analysis 1: Comparison: Period1: PF-07321332 300 mg/Ritonavir 100 mg vs Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.05, Mixed Models Analysis; Specified in comments = 44.50, 90% CI 2-sided [33.77 to 58.65] — Mixed Model was fitted to obtain: 1.Ratio of adjusted geometric means 2.90% CI for the ratios

3. Secondary Outcome: Cmax of Ritonavir
Description: Cmax was defined as maximum observed plasma concentration and can be observed directly from data.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
Number analyzed (Participants) | 12 | 10
ng/mL | 359.3 (46) | 96.07 (71)
Statistical Analysis 1: Comparison: Period1: PF-07321332 300 mg/Ritonavir 100 mg vs Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.05, Mixed Models Analysis; Specified in comments = 25.59, 90% CI 2-sided [18.76 to 34.91] — Mixed Model was fitted to obtain: 1.Ratio of adjusted geometric means 2.90% CI for the ratios

4. Secondary Outcome: AUCinf of Ritonavir
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
Number analyzed (Participants) | 12 | 8
ng*hr/mL | 3599 (47) | 677.6 (61)
Statistical Analysis 1: Comparison: Period1: PF-07321332 300 mg/Ritonavir 100 mg vs Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.05, Mixed Models Analysis; Specified in comments = 16.57, 90% CI 2-sided [13.32 to 20.60] — Mixed Model was fitted to obtain: 1.Ratio of adjusted geometric means 2.90% CI for the ratios

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An Adverse event (AE) was any untoward medical occurrence in a participant. A serious AE was any untoward medical occurrence at any dose that resulted in death; was life-threatening; required hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity, congenital anomaly/birth. An AE was considered treatment-emergent AE (TEAE) if the event occurred during the on-treatment period. A treatment-related AE was any untoward medical occurrence attributed to the study drug in a participant who received study drug. A treatment-related SAE was a treatment-related AE and was defined as any untoward medical occurrence at any dose that: was fatal or life-threatening; resulted in persistent or significant disability/incapacity; constituted a congenital anomaly/birth defect; was medically significant; required inpatient hospitalization or prolongation of existing hospitalization. Relatedness to study drug was assessed by the investigator.
Time Frame: Screening up to Day 3 in Period 1; Day 1 up to 35 days from administration of the final dose of study intervention or early termination/discontinuation in Period 2 (maximum of approximately 12 weeks)
Population: The analysis population included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
Number analyzed (Participants) | 12 | 12
Participants
  Participants with all-causality adverse events | 4 | 9
  Participants with all-causality serious adverse events | 0 | 0
  Participants with treatment related adverse events | 1 | 6
  Participants with treatment related serious adverse events | 0 | 0

6. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Safety laboratory assessments included hematology, urinalysis, and clinical chemistry. All the safety laboratory samples were collected following at least a 4 hour fast.
Time Frame: Screening, Day -1 prior to dosing, and Day 2 in Period 1; Days 3, 6, 9, 12, 16 or early termination/discontinuation in Period 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
Number analyzed (Participants) | 12 | 12
Participants
  Hemoglobin (g/dL) <0.8x lower limit of normal (LLN) | 0 | 1
  Hematocrit (%) <0.8x LLN | 0 | 1
  Erythrocytes (10^6/mm^3) <0.8x LLN | 0 | 1
  Lymphocytes (10^3/mm^3) <0.8x LLN | 0 | 2
  Neutrophils (10^3/mm^3) <0.8x LLN | 0 | 1
  Eosinophils/Leukocytes (%) >1.2x upper limit of normal (ULN) | 1 | 4
  Monocytes/Leukocytes (%) >1.2x ULN | 1 | 5
  Alanine Aminotransferase (U/L) >3.0x ULN | 0 | 4
  Sodium (milliequivalent per liter (mEq/L)) <0.95x LLN | 0 | 1
  Urobilinogen (EU/dL) ≥1 | 0 | 1
  Fibrinogen (mg/dL) >1.25x Baseline | 0 | 1
  URINE Hemoglobin ≥1 | 0 | 3

7. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs including single supine blood pressure and pulse rate were performed following at least a 5 minute rest in a supine position. Blood pressure (BP) and pulse rate (PR) assessments were performed after collection of electrocardiograms (ECGs) and prior to collection of blood draws if planned together. Respiratory rate (RR) was also evaluated.
Time Frame: Screening and Day 1 pre-dose, and at 1.5, 8, and 24 hours post dose in Period 1; Days 2, 3, 4, 6, 8, 10, 12, Day 14 pre-dose, and at 1.5, 8, 24, and 48 hours post-dose or early termination/discontinuation in Period 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
Number analyzed (Participants) | 12 | 12
Participants
  Supine diastolic blood pressure value <50 mmHg | 0 | 0
  Supine diastolic blood pressure change ≥20mmHg increase | 0 | 1
  Supine diastolic blood pressure change ≥20mmHg decrease | 0 | 0
  Supine pulse rate value <40 beats per minute(bpm) | 0 | 0
  Supine pulse rate value >120 bpm | 0 | 0
  Supine systolic blood pressure value <90mmHg | 1 | 0
  Supine systolic blood pressure change ≥30mmHg decrease | 0 | 0
  Supine systolic blood pressure change ≥30mmHg increase | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Change in Electrocardiogram (ECG) Findings
Description: All ECG assessments (triplicate) were made after at least a 10 minute rest in a supine position and prior to any blood draws or vital sign measurements.
Time Frame: Screening and Day 1 pre-dose, and at 1.5, 8, and 24 hours post dose in Period 1; Days 2, 3, 4, Day 14 pre-dose, and at 1.5, 8, 24, and 48 hours post-dose or early termination/discontinuation in Period 2
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
Number analyzed (Participants) | 12 | 12
Participants
  PR interval, aggregate value ≥300 milliseconds (msec) | 0 | 0
  PR interval, aggregate percent change ≥25/50% | 0 | 0
  QRS duration, aggregate value ≥140 msec | 0 | 0
  QRS duration, aggregate percent change ≥50% | 0 | 0
  QTCF interval, aggregate value >450 msec and ≤480 msec | 0 | 0
  QTCF interval, aggregate value >480 msec and ≤500 msec | 0 | 0
  QTCF interval, aggregate value >500 msec | 0 | 0
  QTCF interval, aggregate change ≥30 msec and ≤60 msec | 0 | 0
  QTCF interval, aggregate change >60 msec | 0 | 0

9. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of PF-07321332
Description: Tmax was defined as time to reach maximum observed plasma concentration and can be observed directly from data as time of first occurrence.
Time Frame: as for outcome 1
Population: The pharmacokinetic (PK) parameter analysis population was defined as all participants assigned to investigational product and treated who had at least 1 of the PK parameters of primary interest measured. Number of participants analyzed represents the number of participants contributing to the summary statistics for Tmax.
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
Number analyzed (Participants) | 12 | 10
hour (hr) | 3.00 [1.02 to 6.00] | 1.50 [0.500 to 4.00]

10. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-07321332
Description: AUClast was defined as area under the plasma concentration-time profile from time 0 to the time of last observed quantifiable plasma concentration (Clast) and was determined by Linear/Log trapezoidal method.
Time Frame: as for outcome 1
Population: The analysis population was defined as all participants assigned to investigational product and treated who had at least 1 of the PK parameters of primary interest measured. Number of participants analyzed represents the number of participants contributing to the summary statistics for AUClast.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
Number analyzed (Participants) | 12 | 10
ng*hr/mL | 22450 (23) | 10050 (58)
Statistical Analysis 1: Comparison: Period1: PF-07321332 300 mg/Ritonavir 100 mg vs Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.05, Mixed Models Analysis; Specified in comments = 44.59, 90% CI 2-sided [33.99 to 58.50] — Mixed Model was fitted to obtain: 1.Ratio of adjusted geometric means 2.90% CI for the ratios

11. Secondary Outcome: Apparent Oral Clearance (CL/F) of PF-07321332
Description: CL/F was defined as apparent clearance. Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is a quantitative measure of the rate at which a drug substance is removed from the blood. CL/F is calculated as dose/AUCinf. AUCinf = area under the plasma concentration versus time curve from time zero extrapolated to infinite time.
Time Frame: as for outcome 1
Population: The analysis population was defined as all participants assigned to investigational product and treated who had at least 1 of the PK parameters of primary interest measured. Number of participants analyzed represents the number of participants contributing to the summary statistics for CL/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/hr)
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
Number analyzed (Participants) | 12 | 10
Liter per hour (L/hr) | 13.06 (23) | 29.17 (58)

12. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of PF-07321332
Description: Vz/F was defined as apparent volume of distribution. Vz/F is calculated as Dose/(AUCinf * kel), where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve.
Time Frame: as for outcome 1
Population: The analysis population was defined as all participants assigned to investigational product and treated who had at least 1 of the PK parameters of primary interest measured. Number of participants analyzed represents the number of participants contributing to the summary statistics for Vz/F.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
Number analyzed (Participants) | 12 | 10
Liter (L) | 109.4 (38) | 157.2 (69)

13. Secondary Outcome: Terminal Half-Life ( t1/2) of PF-07321332
Description: t1/2 was defined as the time measured for the plasma concentration of drug to decrease by one half. t1/2 is calculated as Loge(2)/kel, where kel is the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Only those data points judged to describe the terminal log-linear decline was used in the regression.
Time Frame: as for outcome 1
Population: The analysis population was defined as all participants assigned to investigational product and treated who had at least 1 of the PK parameters of primary interest measured. Number of participants analyzed represents the number of participants contributing to the summary statistics for t1/2.
Measure: Mean (Standard Deviation); unit: hours (hr)
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
Number analyzed (Participants) | 12 | 8
hours (hr) | 6.053 (1.7939) | 3.845 (0.99642)

14. Secondary Outcome: Tmax of Ritonavir
Description: as for outcome 9
Time Frame: as for outcome 1
Population: The analysis population was defined as all participants assigned to investigational product and treated who had at least 1 of the PK parameters of primary interest measured. Number of participants analyzed represents the number of participants contributing to the summary statistics for Tmax.
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
Number analyzed (Participants) | 12 | 10
hour (hr) | 3.98 [1.48 to 4.20] | 1.98 [0.983 to 4.00]

15. Secondary Outcome: AUClast of Ritonavir
Description: AUClast was defined as area under the plasma concentration-time profile from time 0 to the time of Clast and was determined by Linear/Log trapezoidal method.
Time Frame: as for outcome 1
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
Number analyzed (Participants) | 12 | 10
ng*hr/mL | 3414 (47) | 466.2 (104)
Statistical Analysis 1: Comparison: Period1: PF-07321332 300 mg/Ritonavir 100 mg vs Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.05, Mixed Models Analysis; Specified in comments = 12.92, 90% CI 2-sided [9.28 to 17.99] — Mixed Model was fitted to obtain: 1.Ratio of adjusted geometric means 2.90% CI for the ratios

16. Secondary Outcome: CL/F of Ritonavir
Description: as for outcome 11
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
Number analyzed (Participants) | 12 | 8
L/hr | 27.78 (48) | 147.6 (61)

17. Secondary Outcome: Vz/F of Ritonavir
Description: as for outcome 12
Time Frame: as for outcome 1
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
Number analyzed (Participants) | 12 | 8
L | 234.0 (36) | 697.5 (51)

18. Secondary Outcome: t1/2 of Ritonavir
Description: as for outcome 13
Time Frame: as for outcome 1
Population: The pharmacokinetic (PK) parameter analysis population was defined as all participants assigned to investigational product and treated who had at least 1 of the PK parameters of primary interest measured. Number of participants analyzed represents the number of participants contributing to the summary statistics for t1/2.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
Number analyzed (Participants) | 12 | 8
hr | 6.149 (2.2413) | 3.345 (0.79964)

ADVERSE EVENTS:
Time Frame: Screening up to Day 3 in Period 1; Day 1 up to 35 days from administration of the final dose of study intervention or early termination/discontinuation in Period 2 (maximum of approximately 12 weeks)
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Period1: PF-07321332 300 mg/Ritonavir 100 mg | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 9/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Period1: PF-07321332 300 mg/Ritonavir 100 mg (N=12) | Period2: Carbamazepine + PF-07321332 300 mg/Ritonavir 100 mg (N=12)
Excessive cerumen production (Ear and labyrinth disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vessel puncture site haematoma (General disorders) | 1 | 1
Asymptomatic COVID-19 (Infections and infestations) | 0 | 1
Transaminases increased (Investigations) | 0 | 5
Altered pitch perception (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 1
Sciatica (Nervous system disorders) | 1 | 0
Poor quality sleep (Psychiatric disorders) | 0 | 1
Polyuria (Renal and urinary disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-07-02): https://cdn.clinicaltrials.gov/large-docs/30/NCT04962230/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/30/NCT04962230/SAP_001.pdf